CLINICAL TRIAL: NCT01359254
Title: Combined Transplantation of Unmanipulated Haploidentical and a SingleCord Blood Unit for Patients With Hematologic Malignancies
Brief Title: Cord Blood Transplantation for Patients With Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: did not accrue enough patients.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-020-B
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Hematological Disease
MeSH Terms: conditions — Hematologic Diseases | interventions — Melphalan; fludarabine; fludarabine phosphate; Antilymphocyte Serum; Busulfan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conditioning Regimen I (Experimental): Arm I contains fludarabine, melphalan, and antithymocyte globulin (ATG)
  Interventions: Drug: Melphalan; Drug: Fludarabine; Drug: Antithymocyte Globulin (ATG)
- Conditioning Regimen II (Experimental): Arm II contains fludarabine, busulfan, antithymocyte globulin (ATG), and total body irradiation (TBI).
  Interventions: Drug: Fludarabine; Drug: Antithymocyte Globulin (ATG); Drug: Busulfan; Drug: Total Body Irradiation (TBI)

INTERVENTIONS:
Drug: Melphalan — Melphalan is given daily for 2 days, overlapping with the completion of fludarabine.
  Other Names: Alkeran; Sarcolysin
  Arms: Conditioning Regimen I
Drug: Fludarabine — Fludarabine is given through the vein daily for 5 days.
  Other Names: fludarabine phosphate; Fludara
Drug: Antithymocyte Globulin (ATG) — ATG is given every other day for 4 days.
Drug: Busulfan — Busulfan is given daily for 4 days.
  Other Names: Myleran; Busulfex IV
  Arms: Conditioning Regimen II
Drug: Total Body Irradiation (TBI) — TBI is given twice on the last day.
  Arms: Conditioning Regimen II

SUMMARY:
The primary objective of this study is to assess the rate of engraftment with combined haploidentical-cord blood transplantation in patients with pre-existing donor specific antibodies and in those with active disease.

DETAILED DESCRIPTION:
Primary Objective

- To assess the rate of engraftment with combined haploidentical-cord blood transplantation in patients with pre-existing donor specific anti-HLA antibodies and in those with active disease

Secondary Objectives

* To determine the long term fate of the haplo transplant and the cord blood transplant in this setting.
* To describe the incidence and severity of acute and chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute leukemia (myeloid or lymphoid)
* Acute leukemia in first remission at high-risk for recurrence
* Chronic myelogenous leukemia in accelerated phase or blast-crisis
* Chronic myelogenous leukemia in chronic phase
* Recurrent or refractory malignant lymphoma or Hodgkin lymphoma
* Chronic lymphocytic leukemia, relapsed or with poor prognostic features
* Multiple myeloma
* Myelodysplastic syndrome
* Chronic myeloproliferative disease
* Hemoglobinopathies
* Aplastic anemia

Exclusion Criteria:

* Zubrod performance status > 2
* Life expectancy is severely limited by concomitant illness
* Patients with severely decreased LVEF or impaired pulmonary function tests
* Estimated Creatinine Clearance <50 ml/min
* Serum bilirubin> 2.0 mg/dl or SGPT >3 x upper limit of normal
* Evidence of chronic active hepatitis or cirrhosis
* HIV-positive
* Patient is pregnant
* Patient or guardian not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine, Melphalan, and ATG: Arm I contains fludarabine, melphalan, and antithymocyte globulin (ATG)
  Melphalan: Melphalan is given daily for 2 days, overlapping with the completion of fludarabine.
  Fludarabine: Fludarabine is given through the vein daily for 5 days.
  Antithymocyte Globulin (ATG): ATG is given every other day for 4 days.
- Fludarabine, Busulfan, ATG, and TBI: Arm II contains fludarabine, busulfan, antithymocyte globulin (ATG), and total body irradiation (TBI).
  Fludarabine: Fludarabine is given through the vein daily for 5 days.
  Antithymocyte Globulin (ATG): ATG is given every other day for 4 days.
  Busulfan: Busulfan is given daily for 4 days.
  Total Body Irradiation (TBI): TBI is given twice on the last day.
Period: Overall Study
Arm/Group | Fludarabine, Melphalan, and ATG | Fludarabine, Busulfan, ATG, and TBI
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fludarabine, Melphalan, and ATG | Fludarabine, Busulfan, ATG, and TBI | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Cord Blood Engraftment by Day 100
Description: Percent of subjects with cord blood engraftment on or before day 100. Detectable cord blood engraftment should be present by day 100 in at least 50% of patients.
  As of 44 days post-transplant, only haploidentical donor chimerism achieved in the one patient enrolled in the Fludarabine, melphalan, and ATG arm. There were no cord cells detected for this patient.
Time Frame: 100 days
Population: The only enrolled patient failed to complete the study due to death.
Arm/Group | Fludarabine, Melphalan, and ATG | Fludarabine, Busulfan, ATG, and TBI
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Survival at Day 100
Description: Percent of subjects who are alive 100 days after the stem cell infusion
Time Frame: 100 days
Population: The only enrolled patient failed to complete the study due to death.
Arm/Group | Fludarabine, Melphalan, and ATG | Fludarabine, Busulfan, ATG, and TBI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Fludarabine, Melphalan, and ATG | Fludarabine, Busulfan, ATG, and TBI
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine, Melphalan, and ATG (N=1) | Fludarabine, Busulfan, ATG, and TBI (N=0)
Septic shock (General disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine, Melphalan, and ATG (N=1) | Fludarabine, Busulfan, ATG, and TBI (N=0)
Acute graft versus host disease (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes